CLINICAL TRIAL: NCT04311658
Title: Safety and Efficacy of the Effect of Isosorbide Mononitrate in Reducing Pain During Levonorgestrel-releasing Intrauterine Device Insertion in Adolescents and Young Women
Brief Title: Safety and Efficacy of the Effect of Isosorbide Mononitrate in Reducing Pain During Levonorgestrel-releasing Intrauterine Device Insertion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: isosorbide mononitrate IUDs
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Contraception
MeSH Terms: interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isosorbide Mononitrate (Experimental): one tablet of Isosorbide Mononitrate (40 mg) vaginally 3 hours prior to LNG-IUD insertion
  Interventions: Drug: Isosorbide Mononitrate 40 MG
- placebo (Placebo Comparator): one tablet of placebo vaginally 3 hours prior to LNG- IUD insertion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isosorbide Mononitrate 40 MG — one tablet of Isosorbide Mononitrate (40 mg) vaginally 3 hours prior to LNG- IUD insertion
  Arms: Isosorbide Mononitrate
Drug: Placebo — one tablet of placebo vaginally 3 hours prior to LNG-IUD insertion
  Arms: placebo

SUMMARY:
the aim of the study is to evaluate the safety and efficacy of isosorbide mononitrate vaginal administration in reducing pain during LNG-IUD insertion in adolescents and young women

ELIGIBILITY:
Inclusion Criteria:

* adolescents and young women requesting LNG-IUD insertion

Exclusion Criteria:

* heavy vaginal bleeding,pregnancy, contraindications to IUD insertion, allergy or contraindication to isosorbide mononitrate, uterine anomaly

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-06-25 (Estimated); Study Completion 2020-07-05 (Estimated)

PRIMARY OUTCOMES:
pain during IUD insertion | 5 minutes
  intensity of patient-perceived pain at time of IUD insertion, using a visual analog scale. The VAS scale is graded from 0 to 10 on a 10 cm horizontal straight line, where
  'zero' corresponds to no pain at all, and '10' to the worst possible pain imaginable.

SECONDARY OUTCOMES:
duration of IUD insertion | 5 minutes
  duration of IUD insertion from speculum in to speculum out in minutes